CLINICAL TRIAL: NCT02074839
Title: A Phase I, Multicenter, Open-Label, Dose-Escalation and Expansion, Safety, Pharmacokinetic, Pharmacodynamic, and Clinical Activity Study of Orally Administered AG-120 in Subjects With Advanced Hematologic Malignancies With an IDH1 Mutation
Brief Title: Study of Orally Administered AG-120 in Subjects With Advanced Hematologic Malignancies With an IDH1 Mutation
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AG120-C-001
Record Dates: First submitted 2014-02-21; First posted 2014-02-28 (Estimated); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Relapsed or Refractory Acute Myeloid Leukemia (AML); Untreated AML; Other IDH1-mutated Positive Hematologic Malignancies; Myelodysplastic Syndromes
Keywords: acute myeloid leukemia; AML; myelodysplastic syndrome; MDS; hematologic malignancies; IDH; Untreated AML; IDH1; relapsed AML; refractory AML
MeSH Terms: conditions — Recurrence; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Hematologic Neoplasms | interventions — ivosidenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AG-120 (Experimental): AG-120 administered continuously as a single agent dosed orally every day of a 28-day cycle.
  Interventions: Drug: AG-120

INTERVENTIONS:
Drug: AG-120 — AG-120 administered continuously as a single agent dosed orally every day of a 28-day cycle. Subjects may continue treatment with AG-120 until disease progression, development of other unacceptable toxicity or hematopoietic stem cell transplant.

SUMMARY:
The purpose of this Phase I, multicenter study is to evaluate the safety, pharmacokinetics, pharmacodynamics and clinical activity of AG-120 in advanced hematologic malignancies that harbor an IDH1 mutation. The first portion of the study is a dose escalation phase where cohorts of patients will receive ascending oral doses of AG-120 to determine maximum tolerated dose (MTD) and/or the recommended Phase II dose. The second portion of the study is a dose expansion phase where four cohorts of patients will receive AG-120 to further evaluate the safety, tolerability, and clinical activity of the recommended Phase II dose. Additionally, the study includes a substudy evaluating the safety and tolerability, clinical activity, pharmacokinetics, and pharmacodynamics of AG-120 in subjects with relapsed or refractory myelodysplastic syndrome with an IDH1 mutation. Anticipated time on study treatment is until disease progression or unacceptable toxicity occurs.

ELIGIBILITY:
Key Inclusion Criteria:

* Subject must be ≥18 years of age.
* Subjects must have documented IDH1 R132 gene-mutated advanced hematologic malignancy based on local or central evaluation.
* Subjects must be amenable to serial bone marrow biopsies, peripheral blood sampling, and urine sampling during the study.
* Subjects must have ECOG PS of 0 to 2.
* Platelet count ≥20,000/µL (Transfusions to achieve this level are allowed).
* Subjects must have adequate hepatic function as evidenced by: Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) ≤3.0 × ULN, unless considered due to leukemic disease and serum total bilirubin ≤1.5 x upper limit of normal (ULN), unless considered due to Gilbert's disease or leukemic disease
* Subjects must have adequate renal function as evidenced by a serum creatinine ≤2.0 × ULN or creatinine clearance >40mL/min based on Cockroft-Gault glomerular filtration rate (GFR)
* Subjects must be recovered from any clinically relevant toxic effects of any prior surgery, radiotherapy, or other therapy intended for the treatment of cancer.
* Female subjects with reproductive potential must have a negative serum pregnancy test within 7 days prior to the start of therapy and on the first day of study drug administration.

Key Exclusion Criteria:

* Subjects who have undergone hematopoietic stem cell transplant (HSCT) within 60 days of the first dose of AG-120, or subjects on immunosuppressive therapy post HSCT at the time of screening, or with clinically significant graft-versus-host disease (GVHD). (The use of a stable dose of oral steroids post HSCT and/or topical for ongoing skin GVHD is permitted.)
* Subjects who received systemic anticancer therapy or radiotherapy <14 days prior to their first day of study drug administration. (Hydroxyurea is allowed prior to enrollment and after the start of AG-120).
* Subjects who received an investigational agent <14 days prior to their first day of study drug administration.
* Subjects who are pregnant or breastfeeding.
* Subjects with an active severe infection or with an unexplained fever >38.5°C during screening visits or on their first day of study drug administration (at the discretion of the Investigator, subjects with tumor fever may be enrolled).
* Subjects with New York Heart Association (NYHA) Class III or IV congestive heart failure or LVEF <40% by echocardiogram (ECHO) or multi-gated acquisition (MUGA) scan within approximately 28 days of C1D1.
* Subjects with a history of myocardial infarction within the last 6 months of screening.
* Subjects with a known unstable or uncontrolled angina pectoris.
* Subjects with a known history of severe and/or uncontrolled ventricular arrhythmias.
* Subjects with known unstable or uncontrolled angina pectoris.
* Subjects with heart-rate corrected QT (QTc) interval ≥450 ms or other factors that increase the risk of QT prolongation or arrhythmic events.
* Patients taking medications that are known to prolong the QT interval
* Subjects with known infection with human immunodeficiency virus (HIV) or active hepatitis B or C.
* Subjects with clinical symptoms suggesting active central nervous system (CNS) leukemia or known CNS leukemia. Evaluation of cerebrospinal fluid is only required if there is a clinical suspicion of CNS involvement by leukemia during screening.
* Subjects with immediately life-threatening, severe complications of leukemia such as uncontrolled bleeding, pneumonia with hypoxia or shock, and/or disseminated intravascular coagulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Estimated)
Dates: Start 2014-03-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Safety/tolerability: incidence of adverse events. | up to 26 weeks, on average
Maximum Tolerated Dose and/or the recommended Phase II dose of AG-120 in subjects with advanced hematologic malignancies. | up to 26 weeks, on average
Assess clinical activity of AG-120 in subjects with relapsed or refractory AML who are enrolled in the Expansion Phase. | up to 26 weeks, on average
Safety/tolerability of treatment with AG-120 in subjects with relapsed or refractory myelodysplastic syndrome. | up to 26 weeks, on average
Assess clinical activity of AG-120 in subjects with relapsed or refractory myelodysplastic syndrome. | up to 26 weeks, on average

SECONDARY OUTCOMES:
Dose Limiting Toxicities of AG-120 in subjects with advanced hematologic malignancies. | up to 26 weeks, on average
Pharmacokinetics of AG-120 in subjects with advanced hematologic malignancies. | up to 26 weeks, on average
  Descriptive statistics will be used to summarize PK parameters for each dose group and, where appropriate, for the entire population. Such parameters will include (but are not limited to) maximum concentration (Cmax), time to maximum concentration (Tmax), AUC, elimination half-life, and the fraction of drug excreted unchanged in the urine.
Pharmacodynamic relationship of AG-120 and 2-HG. | up to 26 weeks, on average
  The potential relationship between plasma exposure of AG-120 and plasma, urine, or bone marrow 2-HG levels will be explored with descriptive and graphical methods.
Clinical Activity of AG-120 in advanced hematologic malignancies according to the 2003 revised IWG criteria for AML or the 2006 modified IWG criteria for MDS or MDS/myeloproliferative neoplasms (MPN). | up to 26 weeks, on average
Serial blood sampling at specified time points for determination of plasma concentration-time profiles and PK parameters (Cmax) of AG-120 in subjects with R/R MDS. | up to 26 weeks, on average
Serial blood sampling at specified time points for determination of plasma concentration-time profiles and PK parameters (Tmax) of AG-120 in subjects with R/R MDS. | up to 26 weeks, on average
Serial blood sampling at specified time points for determination of plasma concentration-time profiles and PK parameters (AUC) of AG-120 in subjects with R/R MDS. | up to 26 weeks, on average
Blood and bone marrow sampling at specified time points for determination of 2-HG levels to characterize the percent of 2-HG inhibition of AG-120 in plasma and bone marrow. | up to 26 weeks, on average

CONTACTS AND LOCATIONS:
Locations (30):
- United States (26):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic-AZ, Phoenix, Arizona
  - City of Hope, Duarte, California
  - University of California-Los Angeles, Los Angeles, California
  - University of California-San Francisco, San Francisco, California
  - University of Colorado Denver, Aurora, Colorado
  - Mayo Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Moffit Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University Medical Hospital, Chicago, Illinois
  - John Hopkins Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Center, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cornell Cancer Center, New York, New York
  - Duke Cancer Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
- France (4):
  - Hopital La Timone, Marseille
  - Hopital Haut-Leveque, Pessac
  - Central Lyon Sud, Pierre-Bénite
  - Institute Gustave Roussly (IGR), Villejuif

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: https://clinicaltrials.servier.com/

REFERENCES:
- [Background] Sun M, Yin Q, Liang Y, Chang C, Zheng J, Li J, Ji C, Qiu H, Li J, Gong Y, Luo S, Zhang Y, Chen R, Shen Z, Yue Z, Wang S, Shi Q, Yang J, Jin J, Wang J. Ivosidenib in Chinese patients with relapsed or refractory isocitrate dehydrogenase 1 mutated acute myeloid leukemia: a registry study. Blood Sci. 2024 Jun 20;6(3):e00196. doi: 10.1097/BS9.0000000000000196. eCollection 2024 Jul. PMID 38911469
- [Derived] DiNardo CD, Roboz GJ, Watts JM, Madanat YF, Prince GT, Baratam P, de Botton S, Stein A, Foran JM, Arellano ML, Sallman DA, Hossain M, Marchione DM, Bai X, Patel PA, Kapsalis SM, Garcia-Manero G, Fathi AT. Final phase 1 substudy results of ivosidenib for patients with mutant IDH1 relapsed/refractory myelodysplastic syndrome. Blood Adv. 2024 Aug 13;8(15):4209-4220. doi: 10.1182/bloodadvances.2023012302. PMID 38640348
- [Derived] Jiang X, Wada R, Poland B, Kleijn HJ, Fan B, Liu G, Liu H, Kapsalis S, Yang H, Le K. Population pharmacokinetic and exposure-response analyses of ivosidenib in patients with IDH1-mutant advanced hematologic malignancies. Clin Transl Sci. 2021 May;14(3):942-953. doi: 10.1111/cts.12959. Epub 2021 Jan 25. PMID 33493392
- [Derived] Choe S, Wang H, DiNardo CD, Stein EM, de Botton S, Roboz GJ, Altman JK, Mims AS, Watts JM, Pollyea DA, Fathi AT, Tallman MS, Kantarjian HM, Stone RM, Quek L, Konteatis Z, Dang L, Nicolay B, Nejad P, Liu G, Zhang V, Liu H, Goldwasser M, Liu W, Marks K, Bowden C, Biller SA, Attar EC, Wu B. Molecular mechanisms mediating relapse following ivosidenib monotherapy in IDH1-mutant relapsed or refractory AML. Blood Adv. 2020 May 12;4(9):1894-1905. doi: 10.1182/bloodadvances.2020001503. PMID 32380538
- [Derived] Fan B, Dai D, DiNardo CD, Stein E, de Botton S, Attar EC, Liu H, Liu G, Lemieux I, Agresta SV, Yang H. Clinical pharmacokinetics and pharmacodynamics of ivosidenib in patients with advanced hematologic malignancies with an IDH1 mutation. Cancer Chemother Pharmacol. 2020 May;85(5):959-968. doi: 10.1007/s00280-020-04064-6. Epub 2020 Apr 15. PMID 32296873
- [Derived] Roboz GJ, DiNardo CD, Stein EM, de Botton S, Mims AS, Prince GT, Altman JK, Arellano ML, Donnellan W, Erba HP, Mannis GN, Pollyea DA, Stein AS, Uy GL, Watts JM, Fathi AT, Kantarjian HM, Tallman MS, Choe S, Dai D, Fan B, Wang H, Zhang V, Yen KE, Kapsalis SM, Hickman D, Liu H, Agresta SV, Wu B, Attar EC, Stone RM. Ivosidenib induces deep durable remissions in patients with newly diagnosed IDH1-mutant acute myeloid leukemia. Blood. 2020 Feb 13;135(7):463-471. doi: 10.1182/blood.2019002140. PMID 31841594
- [Derived] DiNardo CD, Stein EM, de Botton S, Roboz GJ, Altman JK, Mims AS, Swords R, Collins RH, Mannis GN, Pollyea DA, Donnellan W, Fathi AT, Pigneux A, Erba HP, Prince GT, Stein AS, Uy GL, Foran JM, Traer E, Stuart RK, Arellano ML, Slack JL, Sekeres MA, Willekens C, Choe S, Wang H, Zhang V, Yen KE, Kapsalis SM, Yang H, Dai D, Fan B, Goldwasser M, Liu H, Agresta S, Wu B, Attar EC, Tallman MS, Stone RM, Kantarjian HM. Durable Remissions with Ivosidenib in IDH1-Mutated Relapsed or Refractory AML. N Engl J Med. 2018 Jun 21;378(25):2386-2398. doi: 10.1056/NEJMoa1716984. Epub 2018 Jun 2. PMID 29860938
- [Derived] Birendra KC, DiNardo CD. Evidence for Clinical Differentiation and Differentiation Syndrome in Patients With Acute Myeloid Leukemia and IDH1 Mutations Treated With the Targeted Mutant IDH1 Inhibitor, AG-120. Clin Lymphoma Myeloma Leuk. 2016 Aug;16(8):460-5. doi: 10.1016/j.clml.2016.04.006. Epub 2016 May 5. PMID 27245312
- Available data/document: Individual Participant Data Set — https://clinicaltrials.servier.com/
- Available data/document: Study Protocol — https://clinicaltrials.servier.com/
- Available data/document: Statistical Analysis Plan — https://clinicaltrials.servier.com/
- Available data/document: Informed Consent Form — https://clinicaltrials.servier.com/
- Available data/document: Clinical Study Report — https://clinicaltrials.servier.com/
- Available data/document: Study-level clinical trial data — https://clinicaltrials.servier.com/